CLINICAL TRIAL: NCT03141658
Title: A Randomized, Single-blind, Parallel-group Study to Evaluate the Effects of TS-134 on Ketamine-induced BOLD Signals in Resting fMRI in Healthy Adult Subjects
Brief Title: Effects of TS-134 on Ketamine-induced BOLD Signals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TS134-US103
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
Keywords: TS-134; ketamine; fMRI
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TS-134 20 mg (Experimental)
  Interventions: Drug: TS-134; Other: Ketamine
- TS-134 60 mg (Experimental)
  Interventions: Drug: TS-134; Other: Ketamine
- Placebo (Experimental)
  Interventions: Drug: Placebo; Other: Ketamine

INTERVENTIONS:
Drug: TS-134 — Multiple dose titrations from 10 mg to 20 mg once daily for 6 days
  Arms: TS-134 20 mg
Drug: TS-134 — Multiple dose titrations from 10 mg to 60 mg once daily for 6 days
  Arms: TS-134 60 mg
Drug: Placebo — Multiple doses of placebo once daily for 6 days
  Arms: Placebo
Other: Ketamine — 0.23 mg/kg bolus over one minute on Screening (baseline) and Day 6

SUMMARY:
The purpose of this study is to evaluate the effects of TS-134 on ketamine-induced BOLD signals in ROIs in resting fMRI in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects between 18 and 55 years of age inclusive (at the time of initial informed consent)
* Body weight ≥ 45 and ≤ 87 kg
* Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2

Exclusion Criteria:

* Female subjects who are pregnant, intend to become pregnant, or are breastfeeding
* History or presence of psychiatric or neurologic disease or condition
* History of first-degree relative with schizophrenia or mood disorder with psychosis
* History of alcohol or drug abuse
* History of recreational ketamine use, recreational PCP use, or an adverse reaction to ketamine
* History of violence
* Presence or positive history of significant medical illness, including high blood pressure, low blood pressure or orthostatic hypotension
* Any subjects who show subthreshold ketamine BOLD response
* Metal implants, pacemaker, other metal or paramagnetic objects contained within the body
* Claustrophobia
* Subject with any history of suicidal behavior or is currently at risk of suicide in the opinion of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI signals in pre-specified ROIs | Screening and Day 6
  Changes in ketamine-induced BOLD fMRI signals in pre-specified ROIs (anterior cingulate cortex (ACC) and anterior insula) following administrations of TS-134

SECONDARY OUTCOMES:
BOLD fMRI signals in whole brain | Screening and Day 6
  Changes in ketamine-induced BOLD fMRI signals in whole brain following administrations of TS-134
Brief Psychiatric Rating Scale (BPRS) | Screening and Day 6
  Changes in BPRS scores following administrations of TS-134
Clinician Administered Dissociative State Scale (CADSS) | Screening and Day 6
  Changes in CADSS scores following administrations of TS-134

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Lieberman, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No